CLINICAL TRIAL: NCT01827280
Title: Acute and Short-term Chronic Effects of Galvus (Vildagliptin) on Endothelial Function and Oxidative Stress on Recently Diagnosed Type 2 Diabetic Obese Women: the Role of Intestinal Peptides During Lipid Overload
Brief Title: Acute and Short-term Chronic Effects of Galvus (Vildagliptin) in Diabetes Type 2 Obese Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Laboratory for Clinical and Experimental Research on Vascular Biology (Unknown)
Responsible Party: Principal Investigator, Luiz Guilherme Kraemer de Aguiar, Professor, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Galvus_2013; BioVasc_2013 (Registry Identifier: BioVasc_2013)
Record Dates: First submitted 2013-04-02; First posted 2013-04-09 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: 1- Microvascular Function; 2-oxidative Stress; 3-inflammation
Keywords: endothelial function; microvascular function; incretins; diabetes mellitus; postprandial lipemia
MeSH Terms: conditions — Diabetes Mellitus | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin 850mg/pill will be administered at lunch time and dinner time for 30 days
  Interventions: Drug: Vildagliptin
- Vildagliptina (Experimental): Vildagliptin 50mg/pill will be administered at 10 AM and at 6 PM also for 30 days.
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin 50mg/pill will be administered at 10 AM and at 6 PM also for 30 days.
  Other Names: Vildagliptin (galvus)

SUMMARY:
The prevalence of obesity and type 2 diabetes mellitus (T2DM) has increased progressively in the past decades, and consequently, a higher incidence of cardiovascular diseases is observed. As this process develops, the endothelial dysfunction is present at early stages of the atherosclerotic disease. Studies conducted at BioVasc/UERJ show the occurrence of endothelial and microvascular dysfunction in obese carriers, even in the absence of dysglycemia. New concepts indicate the endothelium as a possible therapeutic target, and drugs which act not only on diabetes mellitus pathophysiology but also acting as direct cardiovascular protectors bring new therapeutic possibilities. The dipeptidyl-peptidase-4 inhibitors (DPP4), such as vildagliptin, are drugs used on the T2DM treatment. Its incretin mimetic and insulinotropic effects are already well established and several other studies show its effectiveness in reducing glycated hemoglobin, even in monotherapy.

Currently, fat rich foods are being increasingly introduced in the western way of life and recent evidence suggests that the postprandial lipemia (LPP) is related to cardiovascular risk. A better glucose control using vildagliptin can reduce the oxidative stress, and consequently promote a better microvascular and endothelial reactivity. However, vildagliptin can have an additional cardiovascular protective action, not only because of its effect on glycemia and oxidative stress reduction, but maybe because of its direct effect on intestinal peptides with postprandial lipemia reduction. To test this hypothesis, we will proceed the following exams: venous occlusion pletysmography, nailfold videocapilaroscopy and laser-Doppler flowmetry aiming to evaluate vascular reactivity on muscle and at cutaneous site. Anoter group of patients with the same clinical charactherisitics will use metformin, in order to compare its effects with those obtained from the use of Vildaglitpin. Our purpose is to determine whether vildagliptin, evaluated in obese and diabetic women, has vascular protective effects, and whether the regulatory mechanisms of these actions correlate with oxidative stress, inflammatory markers and intestinal peptides in baseline state and after a lipid overload.

ELIGIBILITY:
Inclusion Criteria:

* All patients should have BMI > 30kg/m²
* Present untreated diabetes mellitus type 2
* Age between 19 and 50 years
* Waist Circumference > 80 cm

Exclusion Criteria:

* Renal, coronary vascular or peripheral, hematologic or hepatic disease
* Presence of severe hypertriglyceridemia (> 400mg/dl)
* Smokers
* Significant body mass loss (> 5%) within the six months prior to the study

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in microcirculation function at 30 days | Before and after 30 days
  For this study, there will be used two methods, the traditional one, which consists in assessing the microcirculation parameters by dynamic nailfold videocapillaroscopy technique carried out in the nailfold pleat of the fourth finger on the left hand.

SECONDARY OUTCOMES:
Change from Baseline in endothelial function at 30 days | before and after 30 days (intervention)
  LDF is a method for continuous non invasive determination of the microvascular perfusion, where the study of cutaneous vasomotion by spectral analysis of Laser Doppler signal allows the exploration of five frequency components: endothelial, myogenic, sympathetic, respiratory and cardiac, involved in answers to the stimuli. Therewith vasomotion during the whole study period will be assessed, to find differences in baseline, 30, 60, 120 and 180 min after the meal rich in lipids.

OTHER OUTCOMES:
Change from Baseline in incretins and inflammation markers at 30 days | basal and after 30 days (intervention)
  Through kits read by Multiplex® appliance, inflammatory markers will be evaluated, all simultaneously, with small sample quantity (from 10 to 50µL).

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for Clinical and Experimental Research on Vascular Biology, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Schiapaccassa A, Maranhao PA, de Souza MDGC, Panazzolo DG, Nogueira Neto JF, Bouskela E, Kraemer-Aguiar LG. 30-days effects of vildagliptin on vascular function, plasma viscosity, inflammation, oxidative stress, and intestinal peptides on drug-naive women with diabetes and obesity: a randomized head-to-head metformin-controlled study. Diabetol Metab Syndr. 2019 Aug 23;11:70. doi: 10.1186/s13098-019-0466-2. eCollection 2019. PMID 31462933